CLINICAL TRIAL: NCT03482752
Title: An Open-label, Non-controlled, Multicentre Clinical Trial of Inhaled Molgramostim in Autoimmune Pulmonary Alveolar Proteinosis Patients
Brief Title: Safety Extension Trial of Inhaled Molgramostim in Autoimmune Pulmonary Alveolar Proteinosis
Acronym: IMPALA-X
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: SAV006-03 was initiated before the evaluation of the IMPALA study (NCT02702180) results. Considering these results and authority advice there would not be adequate efficacy and safety data from SAV006-03 and the study was terminated.
Sponsor: Savara Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAV006-03; 2017-004078-32 (EudraCT Number)
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-01

CONDITIONS: Autoimmune Pulmonary Alveolar Proteinosis
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis, Acquired | interventions — molgramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: Open label, non-controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Molgramostim nebulizer solution (300 μg) (Experimental): Open-label treatment with molgramostim nebulizer solution (300 μg) administered intermittently (repetitive cycles of 7 days of treatment followed by 7 days off-treatment).
  Interventions: Drug: Molgramostim

INTERVENTIONS:
Drug: Molgramostim — 300 µg inhaled molgramostim in cycles of once daily administration for 7 days, then 7 days off treatment.
  Other Names: Recombinant human GM-CSF

SUMMARY:
SAV006-03 is an open-label extension study for participants who had completed the IMPALA study.

At the baseline visit, eligible participants may continue or re-start treatment with 300 µg inhaled molgramostim (recombinant human Granulocyte-Macrophage Colony Stimulating Factor; GM-CSF) administered intermittently in cycles of seven days molgramostim, administered once daily, and seven days off treatment.

Participants will be treated with inhaled molgramostim for up to 36 months.

During the trial, whole lung lavage will be applied as rescue therapy.

ELIGIBILITY:
Inclusion Criteria:

* Completer of the IMPALA trial.
* Females who have been post menopausal for >1 year, or females of child-bearing potential who are not pregnant or lactating and are using acceptable contraceptive methods.
* Males agreeing to use using acceptable contraceptive methods.
* Willing and able to provide signed informed consent.

Exclusion Criteria:

* Treatment with GM-CSF products other than molgramostim nebuliser solution within three months of Baseline.
* Treatment with any investigational medicinal product other than inhaled molgramostim within four weeks of Baseline.
* History of allergic reactions to GM-CSF.
* Connective tissue disease, inflammatory bowel disease or other autoimmune disorder requiring treatment associated with significant immunosuppression, e.g. more than 10 mg/day systemic prednisolone.
* Previous experience of severe and unexplained side effects during aerosol delivery of any kind of medicinal product.
* History of, or present, myeloproliferative disease or leukaemia.
* Apparent pre-existing concurrent pulmonary fibrosis.
* Any other serious medical condition which in the opinion of the investigator would make the subject unsuitable for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bonella, Prof., Principal Investigator — Interstitial and Rare Lung Disease Unit, Ruhrlandklinik University Hospital, Essen, Germany
Locations (13):
- Dept. Of Respiratory Diseases & Allergy, Aarhus, Denmark
- CHU Rennes Hospital Pontchaillou, Service de Pneumologie, Rennes, France
- Germany (4):
  - Ruhrlandklinik Essen Westdeutsches Lungenzentrum am Universitätsklinikum Essen GmbH, Essen
  - Asklepios Fachkliniken München - Gauting Klinik für Pneumologie, Gauting
  - Thoraxklinik am Universitätsklinikum Heidelberg Abteilung für Pneumologie und Beatmungsmedizin, Heidelberg
  - Universitätsklinikum Schleswig-Holstein Zentralklinikum Lübeck Medizinische Klinik III - Pneumologie, Lübeck
- Attikon University Hospital 2nd Pulmonary Department Athens Medical School National and Kapodistrian University of Athens, Athens, Greece
- Rabin Medical Center Institute of Pulomonary Medicine, Tel Aviv, Israel
- S.C. Pneumologia Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
- St. Antonius Hospital, Nieuwegein, Netherlands
- Pavlov first Saint Petersburg State Medical Univerisity, Saint Petersburg, Russia
- Yedikule Pulmonary Diseases and Pulmonary Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)
- Dept. Of Intensive Care Unit Royal Brompton Hospital London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: SAV006-03 was an open-label extension trial for participants who had completed the IMPALA study. Among the 30 clinical sites enrolling participants in IMPALA, 13 sites participated in SAV006-03. First participant was enrolled on 16 April 2018 and last participant completed the study on 14 January 2021.
Period: Overall Study
Arm/Group | Molgramostim Nebulizer Solution (300 μg)
Started | 60
Safety Analysis Set (The safety analysis set included all enrolled participants who were exposed to molgramostim nebulizer solution in SAV006-03.) | 59
Completed (The participants who remained in the study when the study was terminated were classified as early terminators.) | 56
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — 1 participant died 24 days after last dose ie outside the definition of treatment-emergent | 1

BASELINE CHARACTERISTICS:
Arm/Group | Molgramostim Nebulizer Solution (300 μg)
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 54
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  Greece | 4
  Netherlands | 6
  Turkey | 7
  Denmark | 3
  United Kingdom | 4
  Italy | 9
  Israel | 4
  France | 4
  Germany | 12
  Russia | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: The primary objective of this trial was safety assessed by adverse event (AE) reporting. Definitions and reporting procedures for AEs were done according to current regulatory standards. AEs were collected by the investigator by a non-leading question and by reporting events directly observed or spontaneously volunteered by participants. Participants were also encouraged to contact the clinic in between visits if they experienced AEs or had any concerns. Treatment-emergent was defined as events occurring on study drug and up to 7 days after last dose of study drug.
Time Frame: 139 weeks
Population: Safety analysis set.
Measure: Number; unit: events
Arm/Group | Molgramostim Nebulizer Solution (300 μg)
Number analyzed (Participants) | 59
events | 165

2. Primary Outcome: Number of Serious TEAEs
Description: Serious TEAEs were defined as any untoward medicinal occurrence or effect that at any dose:
  * Results in death
  * Is life-threatening
  * Requires hospitalisation or prolongation of existing hospitalisation
  * Results in persistent or significant disability or incapacity
  * Is a congenital abnormality or birth defect
  * May jeopardise the participant or may require medical intervention to prevent one or more of the outcomes listed above (Important Medical Events).
Time Frame: 139 weeks
Population: Safety analysis set.
Measure: Number; unit: events
Arm/Group | Molgramostim Nebulizer Solution (300 μg)
Number analyzed (Participants) | 59
events | 8

3. Primary Outcome: Number of Treatment-emergent Adverse Drug Reactions (ADRs)
Description: All AEs were assessed by the investigator for causality (unlikely, possible, probable, not applicable) according to current regulatory standards. AEs which had a 'possible' or 'probable' causality were classified as ADRs.
Time Frame: 139 weeks
Population: Safety analysis set.
Measure: Number; unit: events
Arm/Group | Molgramostim Nebulizer Solution (300 μg)
Number analyzed (Participants) | 59
events | 3

4. Primary Outcome: Number of TEAEs Leading to Treatment Discontinuation
Time Frame: 139 weeks
Population: Safety analysis set.
Measure: Number; unit: events
Arm/Group | Molgramostim Nebulizer Solution (300 μg)
Number analyzed (Participants) | 59
events | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the baseline visit up to a follow-up telephone call, which occurred 2 weeks after study completion (maximum duration 139 weeks).
Description: AEs were collected by the investigator by a non-leading question and by reporting events directly observed or spontaneously volunteered by participants. Participants were also encouraged to contact the clinic in between visits if they experienced AEs or had any concerns.
Arm/Group | Molgramostim Nebulizer Solution (300 μg)
All-Cause Mortality (participants affected / at risk) | 1/59
Serious Adverse Events (participants affected / at risk) | 8/59
Other Adverse Events (participants affected / at risk) | 38/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Molgramostim Nebulizer Solution (300 μg) (N=59)
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
HIV infection CDC Group IV subgroup A (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Molgramostim Nebulizer Solution (300 μg) (N=59)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Fatigue (General disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Nasopharyngitis (Infections and infestations) | 7 (7)
Respiratory tract infection (Infections and infestations) | 4 (7)
COVID-19 (Infections and infestations) | 4 (4)
Bronchitis (Infections and infestations) | 3 (6)
Pneumonia (Infections and infestations) | 3 (4)

LIMITATIONS AND CAVEATS:
No hypothesis/statistical testing was planned for any of the endpoints of this study but only descriptive statistics were to be used. Efficacy endpoints were secondary endpoints. Due to early study termination, only limited efficacy data were available for evaluation and in general, no firm conclusion based on efficacy data are applicable. No deaths occurred during the study but 1 participant died due to COVID-19 24 days after last dose, i.e. outside the definition of 'treatment-emergent'.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT03482752/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT03482752/SAP_001.pdf